CLINICAL TRIAL: NCT02877940
Title: A Randomized Controlled Trial Comparing Proseal Laryngeal Mask Airway, I-gel Airway and Laryngeal Tube Suction-D in Mechanically Ventilated Patients
Brief Title: Comparison of ProSeal Laryngeal Mask Airway, LTS-D and I-gel in Mechanically Ventilated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government Medical College, Haldwani (Other)
Responsible Party: Principal Investigator, Dr Subhro Mitra, Assistant Professor, Government Medical College, Haldwani
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 203/GMC/IEC/04/2014
Record Dates: First submitted 2016-08-17; First posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Airway Morbidity
Keywords: ProSeal LMA; LTS-D; i-gel

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ProSeal Laryngeal mask airway (Active Comparator): ProSeal will be inserted in mechanically ventilated patients undergoing elective surgeries.
  Interventions: Device: ProSeal Laryngeal mask airway
- Laryngeal Tube Suction- Disposable (Active Comparator): LTS-D will be inserted in mechanically ventilated patients undergoing elective surgeries.
  Interventions: Device: Laryngeal Tube Suction- Disposable
- Group I (Active Comparator): i-gel will be inserted in mechanically ventilated patients undergoing elective surgeries..
  Interventions: Device: i-gel

INTERVENTIONS:
Device: ProSeal Laryngeal mask airway — ProSeal was inserted in mechanically ventilated patients undergoing elective surgeries.
  Arms: ProSeal Laryngeal mask airway
Device: Laryngeal Tube Suction- Disposable — LTS-D was inserted in mechanically ventilated patients undergoing elective surgeries.
  Arms: Laryngeal Tube Suction- Disposable
Device: i-gel — i-gel was inserted in mechanically ventilated patients undergoing elective surgeries.
  Arms: Group I

SUMMARY:
The Aim of the study is to compare the clinical performance of p-LMA, i-gel and LTS-D in terms of the efficacy and safety in anaesthetized patient on Mechanical ventilation undergoing elective surgical procedure.

DETAILED DESCRIPTION:
The study aims to draw a comparison between ProSeal LMA, i-gel and LTS-D supraglottic airway devices in terms of the efficacy and safety in anaesthetised patient on Mechanical ventilation undergoing elective surgical procedure.

Methodology: A prospective randomized control study conducted on 150 patients undergoing elective surgical procedure under general anaesthesia at Dr Sushila Tiwari Hospital and Government medical college, Haldwani.

Following detailed pre-anaesthetic check-up, informed written consent was taken from patient fulfilling the required criteria. Patients were randomly allocated into 3 groups namely Group I (i-gel, n=50), Group P (p-LMA, n=50) and Group L (LTS-D, n=50) by online generated randomization.

Standard general anaesthesia protocol was followed and once adequate depth was achieved i-gel or p-LMA or LTS-D appropriate for weight or / and height was selected and inserted. An effective airway was confirmed and device was fixed from maxilla to maxilla.

The three groups were compared with respect to number of Insertion attempts, ease of insertion of device, time taken for placement of device, airway sealing pressure, ease and number of attempts of gastric tube placement and complications noted if any.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists (ASA) class I/II.
* Age 20-60years of either sex.
* Weight between 40-60 kg of either sex.
* Elective Surgical procedures of duration of 1-1½ hour with no need for endotracheal intubation.

Exclusion Criteria:

* Patient with risk factors for difficult airway. (Mouth opening of <2cm, Mallampati class 4, limited neck extension, history of previous difficult intubation)
* Any known pulmonary and cardiovascular diseases.
* Risk of aspiration. (Full stomach, hiatus hernia, gastro-oesophageal reflex disease, emergency surgery)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2014-12; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of Insertion attempts | 10 mins

SECONDARY OUTCOMES:
Grading of insertion of device by Easy or Difficult | 10 min
  Easy insertion is defined as no resistance to insert in first attempt. Any repeat attempt or resistance to insertion is defined as Difficult.
Time taken for placement of device | 10 min
Airway sealing pressure | 10 min
Number of attempts of gastric tube placement | 20 min
Complication | 120 min

CONTACTS AND LOCATIONS:
Overall Officials: Geeta Bhandari, MD, Principal Investigator — Professor

IPD SHARING:
Plan to Share IPD: No